CLINICAL TRIAL: NCT03341351
Title: Use of the Modified Beef Tongue Model for Teaching Repair of Obstetrical
Brief Title: Use of the Modified Beef Tongue Model for Teaching Repair of Obstetrical Fourth-Degree Laceration to Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Joseph Malek, Instructor/Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-300000074
Record Dates: First submitted 2017-10-26; First posted 2017-11-14 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Fourth Degree Perineal Laceration Involving Anal Mucosa; Obstetric; Injury; Obstetric Labor Complications
Keywords: Fourth-degree laceration; Beef tongue model
MeSH Terms: conditions — Wounds and Injuries; Obstetric Labor Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor performing the objective structured assessment of technical skills will be masked to the intervention of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instructional video (Active Comparator): The modified beef tongue video group will be given an instructional video created using the modified beef tongue model to show anatomy and proper repair of the laceration.
  Interventions: Other: Instructional video
- Instructional workshop (Active Comparator): The group randomized to the modified beef tongue instructional workshop will undergo an interactive workshop using the modified beef tongue model to show anatomy and proper repair of the laceration.
  Interventions: Other: Instructional workshop

INTERVENTIONS:
Other: Instructional video — Instructional video using the modified beef tongue model
  Arms: Instructional video
Other: Instructional workshop — Instructional workshop using the modified beef tongue model.
  Arms: Instructional workshop

SUMMARY:
This is a study evaluating the use of the modified beef tongue model for teaching repair of obstetrical fourth-degree laceration to residents. Participants will be randomized to either an instructional video using the modified beef tongue model or to an instructional workshop using the modified beef tongue model. Primary outcome will be measured as change in technical skills score as measured by change from baseline on a validated objective structured assessment of technical skills (OSTATS) for repair of fourth-degree laceration.

DETAILED DESCRIPTION:
Institutional Review Board approval has been obtained and written informed consent will be obtained prior to initiation of the study. All obstetrics and gynecology residents at the University of Alabama will be eligible for the study.

Eligible residents who desire will be enrolled and consented for the trial. Participants will then complete a short pre-intervention knowledge assessment written test and be asked to rate their confidence level in completing a fourth-degree repair based on a Likert scale. The written test is the same as the one used by Patel et al to evaluate residents' knowledge about fourth-degree laceration repair. The questions are based on Williams's obstetric chapter on episiotomy repair and showed construct validity given a significant difference in scores between postgraduate year (PGY)-1 and PGY-4 residents. Participants will also complete a baseline objective structured assessment of technical skills (OSATS) assessment for repair of fourth-degree obstetric laceration on a commercial anatomical replica, the Sultan Anal Sphincter Trainer (Limbs & Things Inc, Savannah, Georgia). This model comes with a replaceable perineal pad that allows approximately 24 repairs before replacement is necessary. The validated OSATS used will be the assessment described by Siddiqui et al and validated on a surgical model. The repair will be videotaped and then distributed to evaluators who will use the 20 item task specific checklist described by Siddiqui et al. The time taken for the repair will be recorded.

Demographic and baseline data will be collected on the participants including PGY level, number of fourth-degree lacerations performed, whether they have read a textbook regarding fourth-degree laceration repair, whether they have read a journal article regarding fourth-degree laceration repair, whether they have attended a didactic session in pelvic anatomy, and whether they have attended a didactic session on fourth-degree laceration repair.

Participants will then be randomized into two groups. Randomization will be performed using a computer-generated block design so that each group has a balanced number of residents in each postgraduate year training level. One group will be randomized to the modified beef tongue video and one will be randomized to the modified beef tongue instructional workshop. The modified beef tongue video group will be given an instructional video created using the modified beef tongue model to show anatomy and proper repair of the laceration. The group randomized to the modified beef tongue instructional workshop will undergo an interactive workshop using the modified beef tongue model to show anatomy and proper repair of the laceration.

The modified beef tongue for the video and workshop will be prepared according to the model previously described in the literature. The modified model includes beef tripe (small intestine) used for anal mucosa and chicken leg muscles for anal sphincter muscle analogs. The tripe is tunneled through the body of the trimmed beef tongue and sutured like an ostomy to simulate the anal canal. The tongue is incised toward the tripe "anal canal." Chicken leg muscles are tunneled from the incision out to the cut edges of the beef tongue to create anal sphincter muscle analogs.

Following the didactic intervention, participants from each group will be given the written knowledge assessment test again and the objective structured assessment of technical skills (OSATS) for repair of fourth-degree laceration on the commercial anatomical replica again. The time taken for the repair will be recorded. Residents will also be asked to evaluate model realism, ease of use, and satisfaction using a Likert scale. The residents will be asked to assess their confidence again using a Likert scale.

The participants will then be crossed over and those who were initially randomized to the video group will then undergo the instructional workshop and the ones initially in the workshop group will be given the instructional video. Participants will then be asked to rate their overall preference between models on a scale of 1 to 10 with 1 being the video and 10 being the instructional workshop. They will also complete the written knowledge test again.

The results of this trial may help to inform to a cost- and time-efficient manner of instruction on the repair of 3rd and 4th degree lacerations. A weakness is that it is unclear whether this will translate to effectiveness at the time of an actual third- and fourth-degree repair.

ELIGIBILITY:
Inclusion Criteria:

* Residents currently in training program at University of Alabama at Birmingham

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Technical skills score | up to 24 weeks
  The primary outcome will be change in technical skills score measured as change from baseline in a validated objective structured assessment of technical skills (OSATS) for repair of fourth degree obstetric laceration. This OSATS was described by Siddiqui et al and is based on a task-specific checklist for fourth-degree lacerations and has a maximum score of 20 and minimum score of 0. The higher the score the better the performance.

SECONDARY OUTCOMES:
Participant preference | up to 24 weeks
  Participant preference of model between instructional video and instructional workshop. Participants will be asked to rate their overall preference between models on a scale of 1 to 10 with 1 being the video and 10 being the instructional workshop.
Knowledge assessment | up to 24 weeks
  Knowledge assessed by written test performed pre- and post-intervention. The written test is the same as the one used by Patel et al to evaluate residents' knowledge about fourth-degree laceration repair. The questions are based on Williams's obstetric chapter on episiotomy repair. The test has a minimum score of 0 and maximum score of 17 with a higher score indicating better performance.
Participant confidence | up to 24 weeks
  Participant's confidence in fourth-degree laceration repair as measured by change in confidence score from pre- to post-intervention. This is based on the participant's response to a 10 point Likert scale with 1 being not confident and 10 being completely confident.
Time of repair | up to 24 weeks
  Time taken for repair of fourth degree laceration
Ease of use of model | up to 24 weeks
  Ease of use of the model as reported by participants. This is based on the participant's response to a 10 point Likert scale with 1 being not easy and 10 being the easiest.
Satisfaction | up to 24 weeks
  Overall satisfaction of each model as reported by participants. This is based on the participant's response to a 10 point Likert scale with 1 being not satisfied and 10 being completely satisfied.
Model realism | up to 24 weeks
  Model realism as reported by participants. This is based on the participant's response to a 10 point Likert scale with 1 being not realistic and 10 being the most realistic.
Factors associated with higher knowledge scores | up to 24 weeks
  Factors associated with higher knowledge scores (e.g. PGY level, number of prior repairs, prior didactics). The written test is the same as the one used by Patel et al to evaluate residents' knowledge about fourth-degree laceration repair. The questions are based on Williams's obstetric chapter on episiotomy repair. The test has a minimum score of 0 and maximum score of 17 with a higher score indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Malek, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama Birmingham Hospital, Birmingham, Alabama, United States

REFERENCES:
- [Background] Siddiqui NY, Stepp KJ, Lasch SJ, Mangel JM, Wu JM. Objective structured assessment of technical skills for repair of fourth-degree perineal lacerations. Am J Obstet Gynecol. 2008 Dec;199(6):676.e1-6. doi: 10.1016/j.ajog.2008.07.054. PMID 19084100
- [Background] Patel M, LaSala C, Tulikangas P, O'Sullivan DM, Steinberg AC. Use of a beef tongue model and instructional video for teaching residents fourth-degree laceration repair. Int Urogynecol J. 2010 Mar;21(3):353-8. doi: 10.1007/s00192-009-1042-3. PMID 19924368
- [Background] Illston JD, Ballard AC, Ellington DR, Richter HE. Modified Beef Tongue Model for Fourth-Degree Laceration Repair Simulation. Obstet Gynecol. 2017 Mar;129(3):491-496. doi: 10.1097/AOG.0000000000001908. PMID 28178060

DOCUMENTS (2):
  • Informed Consent Form (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT03341351/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03341351/Prot_SAP_001.pdf